CLINICAL TRIAL: NCT05681338
Title: Effect of the Coughing Technique During Subcutaneous Heparin Injection on Pain Severity and Individual Satisfaction
Brief Title: Effect of the Coughing Technique During Subcutaneous Heparin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Dilek Yilmaz, PhD, Bursa Uludag University, Department of Nursing, Uludag University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-6/18
Record Dates: First submitted 2022-12-25; First posted 2023-01-12 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Thyroidectomy; Colon Surgery; Cholecystectomy; Inguinal Hernia
Keywords: subcutaneous heparin injection; coughing technique; pain; individual satisfaction; non-pharmacological method
MeSH Terms: conditions — Hernia, Inguinal; Pain

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The measurements were carried out by the first researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the medium intensity coughing technique (Experimental): Immediately before the subcutaneous heparin injection was given, patients were asked to cough twice at a medium level. After that, they were asked to cough ten seconds later for a second time at the same level, and while they were coughing for the second time, the needle was inserted into the tissue.
  Interventions: Other: the medium intensity coughing technique
- the standard injection technique (No Intervention): During the subcutaneous heparin injection, patients were not asked to perform any action, and the injection was given by the standard technique.

INTERVENTIONS:
Other: the medium intensity coughing technique — The medium intensity coughing technique: Immediately before the subcutaneous LMWH injection was given, patients were asked to cough twice at a medium level. After that, they were asked to cough ten seconds later for a second time at the same level, and while they were coughing for the second time, the needle was inserted into the tissue.
  Arms: the medium intensity coughing technique

SUMMARY:
Objective: to examine the effect of the medium intensity coughing technique during subcutaneous low molecular weight heparin injection on pain severity and individual satisfaction in general surgery patients. Method: a prospective, quasi-experimental study included 100 patients who had prescribed a subcutaneous low molecular weight heparin injection once in 24 hours. Each patient received two injections by the same researcher using standard injection technique with medium intensity coughing technique and only standard injection technique.

DETAILED DESCRIPTION:
Aims and objectives: The aim of this study was to examine the effect on the level of pain severity and satisfaction of patients of the medium intensity coughing technique applied to patients during the administration of subcutaneous low molecular weight heparin (LMWH) injection.

Design: This research was a prospective quasi-experimental study. Methods: It was conducted with 100 patients in the General Surgery Clinic of a university hospital in the Marmara Region of Turkey. Subcutaneous LMWH injections were administered by the same nurse to the outer side of the right and left upper arms by the standard injection technique and the medium intensity coughing technique. Immediately after the subcutaneous LMWH injection was given, a researcher who did not know which injection method had been used asked the patients to evaluate their pain levels by the Visual Analog Scale (VAS) and their satisfaction with the performance of the injection by the Visual Individual Satisfaction Scale (VISS).

ELIGIBILITY:
Inclusion Criteria:

* Participating voluntarily in the study
* Being over the age of 18,
* Having a doctor's prescription for subcutaneous low molecular weight heparin 0.6 mL treatment and not yet having begun treatment.
* Having no coagulation disorder, having no disorder that could affect pain perception, -
* Having no incision, lipodystrophy, or finding of infection at the injection site,
* Having no communication problem

Exclusion Criteria:

* Not wanting to participate in the study, or during the course of the research, wishing to withdraw from the study
* Having any condition which would affect the sensation of pain
* Not being able to agree on a place or time
* Being less than 18 years of age

Ages: 22 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Pain assessed by Visual Analog Scale (VAS) | 2 months
  In evaluating the severity of pain felt by the patients during subcutaneous injections, a 10 cm long vertical VAS was used, on which one end represented no pain, and the other end the worst possible pain. The VAS is a commonly used pain assessment scale in clinical settings. Pain severity measurements were evaluated in millimeters.
"Satisfaction assessed by the Visual Individual Satisfaction Scale (VISS) | 2 months
  During the administration of the injection, an evaluation was made to determine individuals' satisfaction using the Visual Individual Satisfaction Scale, which consisted of a vertical 10 cm scale with "I'm very satisfied" written at one end of it and "I'm not at all satisfied" at the other. The Visual Individual Satisfaction Scale incorporated the characteristics of the well-known Visual Analog Scale (VAS). Satisfaction level measurements were evaluated in millimeters.

SECONDARY OUTCOMES:
Weight | 2 months
  weight in kilograms
Height | 2 months
  height in meters
BMI | 2 months
  BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University Hospital, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yilmaz D, Ayhan D, Yilmaz DU, Duzgun F. Effect of the coughing technique during subcutaneous heparin injection on pain severity and individual satisfaction. Rev Lat Am Enfermagem. 2023 May 15;31:e3923. doi: 10.1590/1518-8345.6504.3923. eCollection 2023. PMID 37194813